CLINICAL TRIAL: NCT02157376
Title: Effect of Intravenous Esomeprazole Versus Cimetidine in Prevention of Stress Ulcer Prophylaxis in Chinese Seriously Ill Patients - a Randomized, Double-blind, Parallel-group Study
Brief Title: Stress Ulcer Prophylaxis of Intravenous Esomeprazole in Chinese Seriously Ill Patients
Acronym: SUP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D961OC00002
Record Dates: First submitted 2014-05-28; First posted 2014-06-06 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Stress Ulcer Prophylaxis
Keywords: SUP; Upper GI bleeding; Seriously ill patients
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Esomeprazole; Cimetidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esomeprazole active treatment (Experimental): iv esomeprazole 30 min intermittent infusions given for maximum 14 days
  Interventions: Drug: Esomeprazole
- Cimetidine active treatment (Active Comparator): iv cimetidine 30 min bolus infusion followed by iv cimetidine continuous infusion given for maximum 14 days
  Interventions: Drug: Cimetidine

INTERVENTIONS:
Drug: Esomeprazole — iv esomeprazole 30 min intermittent infusions given for maximum 14 days
  Other Names: Nexium
  Arms: Esomeprazole active treatment
Drug: Cimetidine — iv cimetidine 30 min bolus infusion followed by iv cimetidine continuous infusion given for maximum 14 days
  Other Names: Tagamet
  Arms: Cimetidine active treatment

SUMMARY:
The efficacy of esomeprazole will be compared versus cimetidine (a drug that previously demonstrated prevention of bleeding events) during treatment period in proportion of patients for the prevention of upper GI bleeding.

DETAILED DESCRIPTION:
Stress related upper Gastrointestinal (GI) bleedings are important events associated with morbidity and mortality among seriously ill patients. Data from the literature suggest that stress ulcer prevention with effective acid suppressive treatment can reduce bleeding events and is thus an important therapy in high-risk patients. Esomeprazole has the potential to reduce gastric acidity for prolonged periods of time adequate for both preventing mucosal damage and facilitating coagulation. This study is to reveal whether intravenous (iv) esomeprazole is effective in preventing upper gastrointestinal bleeding and if it is tolerated by Chinese seriously ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill patients
2. Requirement for mechanical ventilation
3. At least one major risk factor for stress ulcer related bleeding

Exclusion Criteria:

1. History of gastric or oesophageal surgery
2. Evidence of active GI bleeding
3. Advanced renal disease
4. Treatment with any Proton Pump Inhibitors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xinyu Qin, Principal Investigator — Professor and Chairman, Department of General Surgery,Zhongshan,Hospital, Fudan University
Locations (15):
- China (15):
  - Research Site, Baotou
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guilin
  - Research Site, Haikou
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Xi'an
  - Research Site, Zhanjiang

REFERENCES:
- [Derived] Lou W, Xia Y, Xiang P, Zhang L, Yu X, Lim S, Xu M, Zhao L, Rydholm H, Traxler B, Qin X. Prevention of upper gastrointestinal bleeding in critically ill Chinese patients: a randomized, double-blind study evaluating esomeprazole and cimetidine. Curr Med Res Opin. 2018 Aug;34(8):1449-1455. doi: 10.1080/03007995.2018.1464132. Epub 2018 Apr 20. PMID 29638148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 343 patients were enrolled from 27 centres in China. The first patient entered the study on 15 July 2014 and the last patient completed the study on 18 February 2016.
  Of the 343 patients enrolled into the study, 311 (90.7%) patients were randomised to treatment.
Pre-assignment Details: 32 patients were not randomised to treatment due to eligibility criteria not being fulfilled.
Groups:
- Esomeprazole: iv Esomeprazole 40 mg bid 30 min intermittent infusion given for maximum 14 days
- Cimetidine: iv Cimetidine 300 mg 30 min bolus infusion, followed by iv Cimetidine continuous infusion (50 mg/h) given for maximum 14 days
Period: Overall Study
Arm/Group | Esomeprazole | Cimetidine
Started | 155 | 156
Completed | 133 | 138
Not Completed | 22 | 18
Not completed — Death | 10 | 4
Not completed — Eligibility criteria not fulfilled | 0 | 1
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Not treated | 8 | 3
Not completed — Investigator's misjudgement | 1 | 2

BASELINE CHARACTERISTICS:
Population: Among 311 randomised patients, 300 patients received randomised treatment: 147 patients in the esomeprazole treatment group and 153 patients in the cimetidine treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Cimetidine | Total
Number analyzed (Participants) | 147 | 153 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (11.8) | 50.1 (12.4) | 50.4 (12.1)
Age, Customized [Number; unit: participants]
  <65 years | 131 | 132 | 263
  >=65 years | 16 | 21 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 81
  Male | 104 | 115 | 219
Race/Ethnicity, Customized [Number; unit: participants]
  Asian/Chinese | 147 | 153 | 300

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Patients With Clinically Significant Upper-GI Bleeding During the Treatment Evaluation Phase
Description: Criteria for a clinically significant upper GI bleeding as:
  1. Bright red blood per NG or OG tube that did not clear after NG or OG tube adjustment and 5 to 10 minutes of at least 100 ml lavage with room temperature normal saline-or,
  2. Persistent gastroccult- positive coffee ground material
  During IMP treatment Day 1-2:
  Persistent gastroccult- positive coffee ground material for at least eight consecutive hours that did not clear with at least 100 ml of lavage with room temperature normal saline.
  During IMP treatment Day 3-14:
  Persistent gastroccult- positive coffee ground material in at least three consecutive gastric aspirates within 2 to 4 hours (at least 60 ±20 minutes apart), that did not clear with at least 100 ml of lavage with room temperature normal saline.
Time Frame: 1-14 days
Population: Full analysis set (FAS). All randomized patients in whom at least one dose of randomized treatment has been initiated.
Measure: Number; unit: % of participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 147 | 153
% of participants | 2.7 | 4.6
Statistical Analysis 1: Comparison: Esomeprazole vs Cimetidine; Assuming a bleeding percent of 6.3% for the active comparator, a risk reduction of 3.7% for esomeprazole, and a 5% non-inferiority margin, 150 patients per treatment arm will provide 94% power to demonstrate non-inferiority. The null hypothesis is that the bleeding rate for iv esomeprazole 40 mg bid exceeds the rate for iv cimetidine by an amount at least as large as 5%; Test type: Non-Inferiority or Equivalence — If the lower bound of the two-sided 95% confidence interval for the difference is larger than -0.05, the non-inferiority claim will be met; p = 0.393, Pearson's Chi-square; Risk Difference (RD) = 1.9, 95% CI 2-sided [-2.8 to 6.5] — The difference in treatment group percentages is given by Cimetidine minus Esomeprazole

2. Secondary Outcome: Proportion of Patients With Any Overt Upper-GI Bleeding (Significant and Non-significant) During the Treatment Evaluation Phase
Description: Criteria for a significant upper GI bleeding as described in primary outcome measure or,
  Criteria for a non-significant upper GI bleeding as:
  1. Bright red blood per NG or OG tube that clear after NG or OG tube adjustment and 5 to 10 minutes of lavage with room temperature normal saline or,
  2. Persistent gastroccult- positive coffee ground material
     During IMP treatment Day 1-2:
     Persistent gastroccult - positive coffee ground material for at less than eight consecutive hours or that clear with at least 100 ml of lavage with room temperature normal saline.
     During IMP treatment Day 3-14:
     Persistent gastroccult - positive coffee ground material in less than three consecutive gastric aspirates within 2 to 4 hours (at least 60±20 minutes apart), or that clear with at least 100 ml of lavage with room temperature normal saline or,
  3. Any clinical signs of hematemesis or melena or haematochezia judged (by the Investigator) to be from an upper GI source.
Time Frame: 1-14 days
Population: Full analysis set (FAS). All randomized patients in whom at least one dose of randomized treatment has been initiated.
Measure: Number; unit: proportion of participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 147 | 153
proportion of participants | 0.109 | 0.105

ADVERSE EVENTS:
Time Frame: AEs will be collected from the time of the first administration of IMP until the end of follow-up, up to 15 days. SAEs will be collected from signed inform consent until the end of follow-up, up to 15 days.
Arm/Group | Cimetidine | Esomeprazole
Serious Adverse Events (participants affected / at risk) | 12/153 | 14/147
Other Adverse Events (participants affected / at risk) | 88/153 | 85/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cimetidine (N=153) | Esomeprazole (N=147)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 3 (3)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral circulatory failure (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cimetidine (N=153) | Esomeprazole (N=147)
Anaemia (Blood and lymphatic system disorders) | 15 (15) | 13 (13)
Constipation (Gastrointestinal disorders) | 14 (15) | 8 (11)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 (13) | 6 (7)
Pyrexia (General disorders) | 25 (31) | 27 (31)
Hepatic function abnormal (Hepatobiliary disorders) | 10 (10) | 9 (9)
Lung infection (Infections and infestations) | 31 (31) | 28 (28)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (10) | 13 (14)
Hypernatraemia (Metabolism and nutrition disorders) | 7 (7) | 9 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (22) | 25 (28)
Hypoproteinaemia (Metabolism and nutrition disorders) | 9 (9) | 11 (11)
Hypotension (Vascular disorders) | 7 (7) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No